CLINICAL TRIAL: NCT01743092
Title: Meeting the Unique Treatment Needs of Female Gamblers: A Workbook and Webinar Effectiveness Pilot Study
Brief Title: Testing Resources: Manual and Webinar Guided Treatment vs. Manual Guided Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Nigel Turner, Independent Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 153-2012
Record Dates: First submitted 2012-11-02; First posted 2012-12-06 (Estimated); Results first posted 2016-04-01 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-01

CONDITIONS: Pathological Gambling
Keywords: Pathological gambling; treatment; online counselling; webinar; workbook
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tutorial Workbook (Other): Tutorial Workbook Group only receives a Tutorial Workbook Group
  Interventions: Behavioral: Tutuorial workbook
- Tutorial Workbook Group plus webinar (Experimental): Tutorial Workbook Group plus webinar will receive in addition, a webinar as an additional resource.
  Interventions: Behavioral: Webinar; Behavioral: Tutuorial workbook

INTERVENTIONS:
Behavioral: Webinar — Some clients will receive a webinar as part of their treatment.
  Other Names: online discussion
  Arms: Tutorial Workbook Group plus webinar
Behavioral: Tutuorial workbook — A work book about their addiciton

SUMMARY:
Research specific to women's gambling treatment needs is limited but suggests a critical need for women sensitive options and reduced barriers to access. This pilot will test the effectiveness of a Tutorial Workbook (TW) both as a self-help tool and used in combination with a webinar. Ontario women(n=48) over the age of 19, with gambling concerns, will be recruited through flyers, on-line and newspaper ads and randomly assigned to one of two groups: (a) TW or (b) TWW (TW plus Webinar). All will complete questionnaires addressing gambling behaviours, personal history and mood states prior to and after the 12 week study. Groups (a) and (b) will also provide feedback on the TW's content and relevance. Group (b) will, in addition, provide feedback on the Webinar Group. TW and TWW will be valuable additions to current treatments, of special importance to reduce barriers for women. The study will contribute to best practices in developing web-based treatments.

DETAILED DESCRIPTION:
Most gambling specific research involves men yet findings are typically generalized to women, a shortcoming addressed in the literature. Women are underrepresented in treatment. A previous study (Boughton and Brewster, 2002) with 365 Ontario women not in treatment, explored barriers and treatment needs. Many respondents indicated that women-only groups and self-help materials would be of value. Using web-based resources to increase treatment options has merit in a growing technological age. This study will introduce two unique forms of treatment, a women friendly tutorial workbook developed specifically to address issues commonly underlying women's gambling and a webinar based group facilitated by a gambling clinician. Group support has been demonstrated to be highly beneficial for women in reducing isolation and shame. The research will assist in developing Best Practices in the problem gambling field, especially for women, a neglected and vulnerable group.

There are two questions:

1. First, to what extent is the Tutorial Workbook effective by itself as a treatment option in helping women make changes to their gambling.
2. What extent is the addition of the webinar discussion group option an incremental benefit to the participant in helping women make changes to their gambling.

Web based therapy has proven effective in the treatment of addiction and mental health issues but more research is needed to assess its efficacy for problem gambling. Self-help tools have been demonstrated as effective in reducing gambling but no women specific tools are available. Evidence of the effectiveness of the TW and TWW treatment options will reduce barriers for hard to serve populations of women and expand options for clinical programs to meet the needs of women unable to attend face to face programs. The TW attends to the unique issues and treatment/support needs of women with gambling concerns.

Ultimately the TW materials, once fully developed, can be made available to the general public as an online tool, used to assist n providing telephone counselling, individually or in a group (Webinar) format or be made available as a self-help paper based utorial workbook.

ELIGIBILITY:
Inclusion Criteria:

* pathological gamblers
* not currently in formal gambling specific treatment
* English proficiency (reading, writing and speech)
* access to private computer and phone
* sufficient computer skills to engage in webinar
* able to fully commit to time demands of weekly participation

Exclusion Criteria:

* active psychosis
* unstable mood disorders
* emotion dysregulation
* extreme social anxiety
* cognitive challenges in reading
* not proficient in in English (reading, writing and speech)
* suicidal behaviours
* current problems with drugs/ alcohol abuse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-11; Primary Completion 2014-11 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nigel E Turner, Ph.D., Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Problem Gambling Treatment Service, Toronto, Ontario, Canada

REFERENCES:
- See also: Website for the Problem Gambling Institute of Ontario and CAMH's problem gambling service — http://www.problemgambling.ca

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tutorial Workbook | Tutorial Workbook Group Plus Webinar
Started | 33 | 26
Completed | 19 | 11
Not Completed | 14 | 15
Not completed — Lost to Follow-up | 14 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tutorial Workbook | Tutorial Workbook Group Plus Webinar | Total
Number analyzed (Participants) | 33 | 26 | 59
Age, Continuous [Mean (Full Range); unit: years] | 51 [32 to 67] | 56 [28 to 70] | 53 [28 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 26 | 59
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  white / european | 22 | 22 | 44
  other | 11 | 4 | 15
Region of Enrollment [Number; unit: participants]
  Canada | 33 | 26 | 59

OUTCOME MEASURES:

1. Primary Outcome: Perceived Stress Scale
Description: The questionnaire asks the client about their perceived stress. The Perceived Stress Scale (Cohen, S., Kamarck, T., and Mermelstein, R. (1983). A global measure of perceived stress. Journal of Health and Social Behavior, 24, 386-396. December 1983) is a scale developed to measure the degree to which situations in one's life are appraised as stressful. Psychological stress has been defined as the extent to which persons perceive (appraise) that their demands exceed their ability to cope. The PSS has become one of the most widely used psychological instruments for measuring nonspecific perceived stress.
  The scale has ten questions asking respondents to circle a number between 0 and 4. (0 the feelings and thoughts during the last month: 0 = Never 1 = Almost Never 2 = Sometimes 3 = Fairly Often 4 = Very Often. The range of possible score is from 0 to 40. Scores around 13 are considered average. Scores of 20 or higher are considered to be indicative of high stress levels.
Time Frame: 12 weeks
Population: The number of data points in this analysis equals the number who completed the study, minus 2. There were 2 missing data points in this analysis because two people did not complete the questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tutorial Workbook | Tutorial Workbook Group Plus Webinar
Number analyzed (Participants) | 17 | 11
units on a scale | 15.2 (7.9) | 14.5 (7.1)

2. Secondary Outcome: DASS Depression
Description: The Depression, Anxiety and Stress Scale (DASS 21) is a 21 item self-report questionnaire developed by Lovibond, S.H. & Lovibond, P.F. (1995, Manual for the Depression Anxiety Stress Scales, 2nd. Ed., Sydney: Psychology Foundation).
  The range of total scores for each subscale is from 0 to 21. Higher values represent a worse outcome. Depression Normal 0-4 Mild 5-6 Moderate 7-10 Severe 11-13 Extremely Severe 14+ Anxiety Normal 0-3 Mild 4-5 Moderate 6-7 Severe 8-9 Extremely Severe 10+ Stress Normal 0-7 Mild 8-9 Moderate 10-12 Severe 13-16 Extremely Severe 17+
Time Frame: 12 weeks
Population: The number of data points in this analysis equals the number who completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tutorial Workbook | Tutorial Workbook Group Plus Webinar
Number analyzed (Participants) | 19 | 11
units on a scale
  depression | 4.3 (4.2) | 3.5 (6.2)
  anxiety | 3.8 (4.9) | 2.4 (3.3)
  Stress | 3.6 (4.0) | 5.7 (4.9)

ADVERSE EVENTS:
Time Frame: 1 year
Description: No adverse reactions were reported.
Arm/Group | Tutorial Workbook | Tutorial Workbook Group Plus Webinar
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/26
Other Adverse Events (participants affected / at risk) | 0/33 | 0/26

LIMITATIONS AND CAVEATS:
The samples were recruited by advertisements and thus were not a true random sample of the population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No